CLINICAL TRIAL: NCT00846521
Title: Postprandial Glycemia in Association With Vascular Disease in Childhood Obesity
Brief Title: Study of Post-meal Blood Sugar Peaks in Association With Vascular Disease in Childhood Obesity
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0603001202; 5K23DK74439-3; 5K23DK074439 (NIH)
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Pediatric Obesity; Insulin Resistance; Impaired Glucose Tolerance; Cardiovascular Disease
Keywords: Pediatric Obesity; Insulin Resistance; Glucose Tolerance; Adolescents; Acarbose; Continuous Glucose Monitoring (CGMS); Endothelial Dysfunction
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Glucose Intolerance; Cardiovascular Diseases | interventions — Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acarbose (Experimental): At baseline, subjects underwent an OGTT and 72 hr of out-patient continuous glucose monitoring. They were treated with acarbose (50 mg with meals three times daily) for 6 weeks and repeat 72 hr CGMS profiles were obtained at the end of the study.
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Acarbose — At baseline, subjects underwent an OGTT and 72 hr of out-patient continuous glucose monitoring. They were treated with acarbose (50 mg with meals three times daily) for 6 weeks and repeat 72 hr CGMS profiles were obtained at the end of the study.
  Other Names: Precose

SUMMARY:
The main purpose of this study is to determine whether treatment with acarbose attenuates post-prandial glycemic excursions in non-diabetic/pre-diabetic obese children as determined by continuous glucose monitoring systems (CGMS). To this effect the current pilot study involves a 6 week intervention with acarbose given to all subjects with either impaired glucose tolerance or an area under the curve of >130 mg/dl during the screening oral glucose tolerance test. Three consecutive days of CGMS are then compared to before and during the intervention. The secondary objective addressed in this protocol is the collection of baseline measures of endothelial function in obese and lean children. Even though the duration of acarbose treatment may be too short to demonstrate a vascular effect, the pre and post intervention data would serve as preliminary data for anticipated future studies that assess the vascular effect of reduced post-prandial blood glucose levels.

DETAILED DESCRIPTION:
We are particularly interested in examining whether acarbose lowered the percentage of glucose excursions ≥ 140 mg/dl in a real-life, home environment. At baseline, subjects underwent an oral glucose tolerance test (OGTT) and 72 hr of out-patient continuous glucose monitoring. They were treated with acarbose (50 mg with meals three times daily) for 6 weeks and repeat 72 hr CGMS profiles were obtained at the end of the study.

ELIGIBILITY:
Obese Subjects:

Inclusion Criteria:

* Obesity (BMI > 97%tile for age and sex matched normative data)
* Good general health, taking no medication on a chronic basis
* Age 12-19 yrs, in puberty (girls: breast: Tanner stage II to V, boys: testicular volume >6ml)
* Girls who are sexually active must use adequate birth control methods(such as barrier method or oral contraception) and must have a negative pregnancy test
* Normal liver function tests

Exclusion Criteria:

* Raynaud's syndrome
* Pregnancy or breastfeeding mothers
* Smokers
* Anemia (Hct < 35)
* Baseline creatinine > 1.0 mg
* Abnormal liver transaminases > 1.5X the upper limit of normal
* Presence of endocrinopathies (Cushing syndrome, hypothyroidism)
* Presence or history of gastrointestinal disorders (Inflammatory bowl disease, irritable bowl disease, hernia, ileus)
* Presence of significant chronic illness of any kind
* Drug therapy (examples of commonly occurring drug therapy include any drugs to treat asthma, hypertension, dyslipidemia, insulin resistance, depression)
* Psychiatric disorders
* History of substance abuse (including anorexic agents)

Control Subjects:

Inclusion Criteria:

* Lean (BMI < 85%tile for age and sex matched normative data)
* Good general health, taking no medication on a chronic basis
* Age 12-25 yrs, in puberty (girls: breast: Tanner stage II to V, boys: testicular volume >6ml)
* Girls who are sexually active must use adequate birth control methods (such as barrier method or oral contraception) and must have a negative pregnancy test

Exclusion Criteria:

* Raynaud's syndrome
* Pregnancy or breastfeeding mothers
* Smokers
* Presence of endocrinopathies (Cushing syndrome, hypothyroidism Presence of significant chronic illness of any kind
* Drug therapy (examples of commonly occurring drug therapy include any drugs to treat asthma, dyslipidemia, hypertension, depression)
* Psychiatric disorders
* History of substance abuse
* First degree relative with either T1DM or T2DM
* Presence of acanthosis nigricans

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tania S Burgert, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acarbose Administration: Acarbose : Subjects assigned to treatment will receive an exact supply of Acarbose to cover the initial 5 weeks of intervention. The medication will be distributed by the investigational pharmacy. Subjects will be instructed on the dosing schedule as follows (due to potential gastrointestinal side effects, the dose will be increased incrementally to desired levels).
  Tablets (dose) of acarbose: Week 1 - 25 mg once a day (with dinner); Week 2 - 50 mg once a day (with dinner); Week 3 - 25 mg with breakfast and 50 mg with dinner; Week 4 - 50 mg with breakfast, 25 mg with lunch and 50 mg with dinner; Week 5-7 - 50 mg with breakfast, 50 mg with lunch and 50 mg with dinner.
Period: Overall Study
Arm/Group | Acarbose Administration
Started | 23
Completed | 12
Not Completed | 11
Not completed — Withdrawal by Subject | 5
Not completed — Did not meet OGTT/ CGMS criteria | 5
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis was only done on subjects who completed the study
Arm/Group | Acarbose Administration
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Glucose Values ≥ 140 mg/dl Over 72 Hours of Glucose Readings Measured With a Continuous Glucose Monitor
Time Frame: At baseline (before treatment)
Population: The number of participants who completed the study were analyzed
Measure: Mean (Standard Deviation); unit: percentage of glucose excursions ≥ 140
Groups:
- Acarbose Administration: At baseline, subjects underwent an OGTT and 72 hr of out-patient continuous glucose monitoring. They were treated with acarbose (50 mg with meals three times daily) for 6 weeks and repeat 72 hr CGMS profiles were obtained at the end of the study
Arm/Group | Acarbose Administration
Number analyzed (Participants) | 12
percentage of glucose excursions ≥ 140 | 8 (8)

2. Primary Outcome: Mean Percentage of Glucose Values ≥ 140 mg/dl Over 72 Hours of Glucose Readings Measured With a Continuous Glucose Monitor
Time Frame: After 6 Weeks (post treatment)
Population: The number of participants who completed the study were analyzed
Measure: Mean (Standard Deviation); unit: percentage of glucose excursions ≥ 140
Arm/Group | Acarbose Administration
Number analyzed (Participants) | 12
percentage of glucose excursions ≥ 140 | 2 (5)

ADVERSE EVENTS:
Arm/Group | Acarbose Administration
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes